CLINICAL TRIAL: NCT03676478
Title: Assessing the Influence of Timing of Enteral Feeding Support in Esophageal Cancer Patients on Muscle functTion and Survival
Brief Title: Assessing Timing of Enteral Feeding Support in Esophageal Cancer Patients on Muscle functTion and Survival
Acronym: EFECTS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: halted prematurely due to futility finding at te occasion of an unplanned interm analysis at 200 participants
Sponsor: University Hospital, Gasthuisberg (Other)
Collaborators: Research Foundation Flanders (Other); Kom Op Tegen Kanker (Other); KU Leuven (Other)
Responsible Party: Principal Investigator, Hans Van Veer, MD, MD, FEBS-OGS, University Hospital, Gasthuisberg
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S61665; 2018-002891-41 (EudraCT Number); 116000000382 (Other Grant/Funding Number: Kom op tegen Kanker (Stand up to Cancer)); T002018N (Other Grant/Funding Number: FWO (Fund for Scientific Research Flanders))
Record Dates: First submitted 2018-07-18; First posted 2018-09-18 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Esophageal Cancer; Nutrition Aspect of Cancer; Postoperative Complications; Muscle Weakness; Sarcopenia; Jejunostomy; Complications
MeSH Terms: conditions — Esophageal Neoplasms; Postoperative Complications; Muscle Weakness; Sarcopenia | interventions — Caloric Restriction

STUDY DESIGN:
Intervention Model Description: Single blinded (for outcome), open label, prospective, randomized, controlled, parallel-group designed interventional study
Who Masked: Outcomes Assessor
Masking Description: The study is single blinded at the level of outcome assessment. As in the postoperative setting it will be clear which subject is in the delayed enteral feeding group, masking cannot be performed for participants, care providers and the investigators. Therefore the study is considered to be open label, but single blinded for the primary outcome analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- start enteral support @ POD1 (No Intervention): The standard of care (SoC) in our department consists of enteral nutritional support of maximum 1000 kilocalories (kCal) through a peroperatively placed jejunostomy feeding tube started at POD 1. Oral caloric intake is resumed at POD 4.
- delayed start enteral support @ POD5 (Active Comparator): As study intervention (INT), a period of caloric restriction is set by starting the enteral nutritional support later, at POD 5. Oral caloric intake is resumed at POD 4, similarly as in the control group. This intervention results in a relative caloric defect of more than 4.000 kCal in the immediate postoperative course.
  Interventions: Other: delayed start enteral support @ POD5

INTERVENTIONS:
Other: delayed start enteral support @ POD5 — instead of caloric suppletion, participants will receive mls of water over the jejunostomy feeding tube daily equivalent to the rate of increase of infusion of the control group as to preserve the same amount of fluid administration through the GI route as the control group.
  This is continued until POD5 12.00h when enteral feeding is started according to the incremental regimen as defined for the SOC group. During the intervention, water is used as to maximize stimulation of the enteral route, however without giving nutritional support and need to prolong iv-infusion for maintaining the fluid balance in the participants. Also subjects in this interventional arm will end up with a caloric suppletion of 1.000kCal/24h by the end of postoperative day 7.
  Other Names: delayed start / caloric restriction
  Arms: delayed start enteral support @ POD5

SUMMARY:
The surgical stress of an esophagectomy causes a detrimental impact on the physiological response of the body. In this perspective, one could question whether the current feeding regimens of starting early nutritional support at postoperative day (POD) 1 have a similar negative impact on the muscle mass as documented in critically ill patients.

This study will introduce relative starvation in the early days following esophagectomy compared to the current regimen of early enteral nutritional support.

The research team aims to investigate whether the negative impact on muscle mass and muscle function might be reduced, which should result in enhanced postoperative recovery. The final result of the study will be a well-documented and scientifically substantiated nutritional regimen for patients who underwent an esophagectomy for cancer.

DETAILED DESCRIPTION:
Patients suffering from oesophageal cancer are known to suffer from important weight loss preoperatively, due to dysphagia attributed to the growing tumour. Postoperatively, the challenge of maintaining weight is even more important given the new way of eating through the gastric conduit that replaces the oesophagus. They often also need to tackle dysphagia caused by an anastomotic stricture and overcome the physiological stress of the operation. As a consequence, almost all patients are confronted with postoperative weight loss. Obviously, patients with a low preoperative weight do not have a lot of reserve and are thus even more at risk of becoming anorectic in the postoperative setting.

This postoperative weight loss has a direct relationship with impaired survival. Therefore, reversing or at least stabilizing the postoperative weight loss might improve survival. The link between weight loss and impaired survival is found in the concept of sarcopenia, the breakdown of muscle fibers. Indeed, by losing muscle strength, patients become too weak for general tasks like bathing, putting clothes on or shopping. In a more pronounced stage, loss of muscle mass is responsible for impaired recovery and eg. the inability to fight against respiratory infections due to lack of cough power.

A logical reaction would therefore be to maximize caloric intake in the peri- and postoperative setting. One could therefore implement extra caloric intake as early as possible in the postoperative track in order to improve recovery. This has been up to now been advocated by scientific organisations like ESPEN (European Society for Clinical Nutrition and Metabolism) by spreading their guidelines on postoperative nutrition.

In contrast, within the field of intensive care and nutrition, discussion has risen about timing of feeding. The focus here shifted in the direction of postponing nutrition to a later stage in the recovery of a sick patient, rather than initiate feeding too soon. Through fundamental research, the concept of impaired autophagy at muscular level in case of early feeding was put forward as underlying mechanism. Muscle cells get swollen and their interlinking structure gets disturbed, resulting in decreased function. The muscle loss itself is triggered by the initial inflammatory storm that these patients go through when their lives are at stake at admission on the ICU. Early energy suppletion seems to aggravate this process even more. This cascade negatively influences recovery. This finding led in our own institution to postpone feeding of patients at the ICU until one week after admission, in order to minimize muscle tissue loss.

The investigators consider the experience in ICU patients as a proof of concept of the postoperative aggravation of sarcopenia in esophageal cancer patients. As patients following esophagectomy are also confronted with a similar catecholamin storm and insulin resistance, they could also be considered to suffer from similar processes that inhibit recovery as patients at the ICU.

The main research hypothesis is therefore that relative energy restriction following surgery would result in better qualitative muscle tissue, in comparison to patients that receive early enteral nutritional support. By doing so, the researchers assume to minimize autophagy at muscular level, resulting in better function and ultimately also in better postoperative recovery. Ultimately, this limitation of muscle loss most likely will have a beneficial effect on survival.

The primary outcome parameter, improvement of muscle function, will be assessed by means of a 6 minute walk test. Apart from this test, several side measurements will be performed - a nutrition diary, activity assessment by means of a MoveMonitor sensor, bio-impedance measurement, quantitive evaluation of muscle mass by CT, qualitative evaluation of muscle quality by muscle biopsy, quality-of-life-questionnaires and continous monitoring of glucose levels during enteral feeding will give the researchers more insight in the underliying mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* Candidates for surgical resection with a curative intent, admitted to our Department.
* Able to understand the study information in Dutch or French and tasks related to the study measurements provided by the researchers.
* Able to consent.
* Patients with cancer of the gastroesophageal junction (GEJ), distal, mid- and proximal thoracic esophagus.
* Patients with early as well as advanced clinical stage esophageal cancer: from clinical stages cT1N0 over cT2+ N+ or cT3 Nx after neo-adjuvant therapy or at the time of staging as a candidate for primary surgery.
* Histology preop: Squamous or adenocarcinoma.
* Patients must undergo at least two-field lymphadenectomy; three-field lymphadenectomy if deemed necessary by the clinical team is not a contraindication for inclusion.
* All access: (robotic assisted) minimal invasive (thoracoscopy & laparoscopy) approach, left thoraco-abdominal incision, hybrid esophageal resection or R thoracotomy + laparotomy
* Partial or subtotal esophagectomy.
* Reconstruction by gastric conduit.
* All anastomoses (intrathoracic or cervical).
* Women of child bearing age with esophageal cancer can be included.

Exclusion Criteria:

* Patients in a definitive chemoradiation protocol, or undergoing rescue resection following definitive chemoradiotherapy.
* Patients expected to die within 12 hours (=moribund patients).
* Patients transferred from another institute after esophageal resection with an established nutritional therapy.
* Patients with a cT4b tumor after neo-adjuvant therapy.
* Patients who are at the time of surgery deemed unresectable or found to be unresectable during surgery.
* Patients with a R2-resection.
* Patients with metastasis at the time of clinical staging.
* Patients undergoing transhiatal resection of the esophagus.
* Patients undergoing total gastrectomy
* Patients undergoing an esophageal resection or esophageal bypass as palliative treatment
* Patients with tumors in the cervical esophagus with a distance less than 3cm from the cricopharyngeal sphincter.
* Patients with pharyngeal cancer undergoing (laryngo-)pharyngectomy with gastric pull-up
* Need for colonic or jejunal interposition
* Patients with a second synchronous malignancy
* Patients with inflammatory bowel disease (as this might interfere with caloric uptake in the small bowel)
* Patients with contra-indications for enteral nutrition.
* Patients already participating in a study with a nutritional intervention.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 239 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2025-05-25 (Actual); Study Completion 2025-12-02 (Actual)

PRIMARY OUTCOMES:
Functional recovery (6mWD - 6-minute Walked Distance) | 5±1 weeks postoperative
  detect a difference in walked distance evaluated by means of a 6-minute walk test

SECONDARY OUTCOMES:
Days alive outside hospital | 90 days postoperative
  number of days alive outside hospital from randomisation until POD90, divided by the number of postoperative days excludng admission days for perioperative chemotherapy (max: 90 days)
Global Health status score | 5+/-1 week postoperative
  General Health Related Quality of Life evaluated by means of participant responses on the European Organisation for Research on the Treatment of Cancer (EORTC) Quality of Life Questionnaire for Cancer QLQ-C30 (generic cancer questionnaire) and Quality of Life Questionnaire QLQ-OES18 (oesophageal cancer disease-specific questionnaire, as an adjoint to the more generic cancer cancer questionnaire).
  Scores are expressed in 4-point Likert scales from 1 to 4; higher score equals worser outcomes.

OTHER OUTCOMES:
Occurrence of readmission | assessed upto 1 year postoperative
  number of readmissions following primary discharge
Variation in 6-minute walked distance | discharge and 90 days postoperative
  Changes in 6-minute walked distances at further time points than the primary parameter
90-day mortality | 90 days postoperative
  status dead or alive following surgery
Overall survival | from operation until 1 year postoperative
  status dead or alive following surgery, after ongoing follow-up for one year
Complications following esophagectomy | assessed upto 1 year postoperative
  complications as defined by the Esophagectomy Complications Consensus Group (ECCG)
Length of hospital stay | from day of operation until hospital discharge after esophagectomy, assessed up to 250 days
  duration of admission, from day of operation until discharge, expressed in days
Reasons for readmission | from operation, assessed upto 1 year postoperative
  Reasons for readmissions following primary discharge, based on the complications list as defined by the Esophagectomy Complications Consensus Group (ECCG)
Quality of life - Patient Reported Outcome Measurement - EORTC QLQ-C30 | from inclusion until 1 year postoperative, every 3 months
  quality of life, assessed by the European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire QLQ-C30, probing quality of life in cancer patients by means of 30 questions - Likert Scales [range 1 to 4, lower is better]
Quality of life - Patient Reported Outcome Measurement - EORTC QLQ-OES18 | from inclusion until 1 year postoperative, every 3 months
  quality of life, assessed by the European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire QLQ-OES18, probing quality of life in oesaphageal cancer patients by means of 18 questions, being more disease specific than the QLQ-C30 questionnaire - Likert Scales [range 1 to 4, lower is better]
Activity levels - Metabolic Equivalents of Tasks (MET) >3 | From inclusion until 3 months postoperative
  monitored by means of a Dynaport® accelerometer; duration per assessment period a subject has performed physical activity with a Metabolic Equivalent of Tasks (MET) greater than >3.
  MET is a measure for energy expenditure with MET >3 corresponding to activity more than sedentary state (MET 0 to 3); higher scores means more active.
Activity related energy expenditure | From inclusion until 3 months postoperative
  monitored by means of a Dynaport® accelerometer, expressed in kCal
Body composition - skeletal muscle mass | From inclusion until 3 months postoperative
  analysis of body composition by means of Seca Body Composition Analyzer 515. Assessed parameter: skeletal muscle mass, expressed in percentage of body weight
Body composition - total body water | From inclusion until 3 months postoperative
  analysis of body composition by means of Seca Body Composition Analyzer 515. Assessed parameter: total body water, expressed in percentage of body weight
Body composition - total body fat | From inclusion until 3 months postoperative
  analysis of body composition by means of Seca Body Composition Analyzer 515. Assessed parameter: total body fat, expressed in percentage of body weight
Body composition - phase angle | From inclusion until 3 months postoperative
  analysis of body composition by means of Seca Body Composition Analyzer 515. Assessed parameter: phase angle, expressed in ° (degrees)
Subcutaneous continuous glycaemia levels in range | baseline measurement for 10 days (preoperative), from POD0 until 10 days postoperative, 10 days following discharge (between POD8-14 on average), 10 days after stop nutritional support
  effect of permissive caloric restriction in the intervention group (detection of eventual hypoglycaemia) and the effect of nocturnal enteral nutrition on the glucose homeostasis in the whole patient cohort - by means of a flash glucose monitoring system (Freestyle, Abbott).
  • total time of 'glycaemia level in range', defined as time with (interstitial) glycaemia level between 70mg/dl and 180mg/dl, expressed in total time (minutes/24h)
Subcutaneous continuous glycaemia levels in hypoglycaemia range | baseline measurement for 10 days (preoperative), from POD0 until 10 days postoperative, 10 days following discharge (between POD8-14 on average), 10 days after stop nutritional support
  effect of permissive caloric restriction in the intervention group (detection of eventual hypoglycaemia) and the effect of nocturnal enteral nutrition on the glucose homeostasis in the whole patient cohort - by means of a flash glucose monitoring system (Freestyle, Abbott).
  • total time of hypoglycaemia, defined as time with interstitial glycaemia level < 70mg/dl, expressed in total time (minutes/24h);
Subcutaneous continuous glycaemia levels in hyperglycaemia range during nocturnal enteral nutrition | baseline measurement for 10 days (preoperative), from POD0 until 10 days postoperative, 10 days following discharge (between POD8-14 on average), 10 days after stop nutritional support
  effect of permissive caloric restriction in the intervention group (detection of eventual hypoglycaemia) and the effect of nocturnal enteral nutrition on the glucose homeostasis in the whole patient cohort - by means of a flash glucose monitoring system (Freestyle, Abbott).
  • total time of hyperglycaemia, defined as time with interstitial glycaemia level > 250mg/dl) during nocturnal enteral feeding between 08 pm and 08 am, expressed in total time (minutes/12h)
Assessment of muscle mass quantity | pre-operative vs. 3 months postoperative
  estimation of muscle quantity/sarcopenia via pre- and postoperative available CT-imaging, in comparing mm² of muscle surface area on L3-level image slice
Assesment of muscle mass quality | biopsy preop, biopsy immediately postintervention (POD8±2 days) and biopsy 5 weeks postop
  microscopic evaluation and assessment of muscle tissue through muscle biopsy; for seperate consented participants only
Complications related to feeding catheter | From date of randomization until the date of removal of catheter, assessed up to 12 months
  recording of infections, luxations, blockages and reasons for reintervention/replacement/reinsertion
Body Mass Index | from inclusion until 3 months postoperative
  weight and height will be combined to report BMI in kg/m^2
Assessment of nutritional and caloric intake | From inclusion until 90 days postoperative
  recording of total caloric intake, proteins and fat (oral intake and administered enteral nutritional support though feeding tube), expressed in kCal, g proteins, g fats, based on feeding diaries (home) and food platter pictures (hospital)
Satiety hormone levels - Incretins: GIP | From inclusion until 90 days postoperative
  Level of variation of satiety hormones between groups, which could influence appetite and weight loss, expressed in pmol/l
Satiety hormone levels - Incretins: GLP-1 | From inclusion until 90 days postoperative
  Level of variation of satiety hormones between groups, which could influence appetite and weight loss, expressed in pmol/l
Levels of fasting blood glycaemia | From inclusion until 90 days postoperative
  Assessment of blood glycaemic profile over the course of the study, at sober state of participant, expressed in mg/dl
Levels of Haemoglobin A1c (HbA1c) | From inclusion until 90 days postoperative
  Assessment of HbA1c profile over the course of the study, at sober state of participant, expressed in percent

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Nafteux, MD, PhD, Study Chair — Department of Thoracic Surgery; Lieven P Depypere, MD, PhD, Principal Investigator — Department of Thoracic Surgery; Michaël Casaer, MD, PhD, Study Chair — Department of Intensive Care Medicine; Hans GL Van Veer, MD, Study Director — Department of Thoracic Surgery
Locations (1):
- University Hospitals Leuven, dept. of Thoracic Surgery, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Van Veer H, Moons J, Darling G, Lerut T, Coosemans W, Waddell T, De Leyn P, Nafteux P. Validation of a new approach for mortality risk assessment in oesophagectomy for cancer based on age- and gender-corrected body mass index. Eur J Cardiothorac Surg. 2015 Oct;48(4):600-7. doi: 10.1093/ejcts/ezu503. Epub 2015 Jan 5. PMID 25564215
- [Background] Casaer MP, Mesotten D, Hermans G, Wouters PJ, Schetz M, Meyfroidt G, Van Cromphaut S, Ingels C, Meersseman P, Muller J, Vlasselaers D, Debaveye Y, Desmet L, Dubois J, Van Assche A, Vanderheyden S, Wilmer A, Van den Berghe G. Early versus late parenteral nutrition in critically ill adults. N Engl J Med. 2011 Aug 11;365(6):506-17. doi: 10.1056/NEJMoa1102662. Epub 2011 Jun 29. PMID 21714640
- [Background] Willcutts KF, Chung MC, Erenberg CL, Finn KL, Schirmer BD, Byham-Gray LD. Early Oral Feeding as Compared With Traditional Timing of Oral Feeding After Upper Gastrointestinal Surgery: A Systematic Review and Meta-analysis. Ann Surg. 2016 Jul;264(1):54-63. doi: 10.1097/SLA.0000000000001644. PMID 26779983
- [Background] Low DE, Alderson D, Cecconello I, Chang AC, Darling GE, D'Journo XB, Griffin SM, Holscher AH, Hofstetter WL, Jobe BA, Kitagawa Y, Kucharczuk JC, Law SY, Lerut TE, Maynard N, Pera M, Peters JH, Pramesh CS, Reynolds JV, Smithers BM, van Lanschot JJ. International Consensus on Standardization of Data Collection for Complications Associated With Esophagectomy: Esophagectomy Complications Consensus Group (ECCG). Ann Surg. 2015 Aug;262(2):286-94. doi: 10.1097/SLA.0000000000001098. PMID 25607756
- [Background] Rabinovich RA, Louvaris Z, Raste Y, Langer D, Van Remoortel H, Giavedoni S, Burtin C, Regueiro EM, Vogiatzis I, Hopkinson NS, Polkey MI, Wilson FJ, Macnee W, Westerterp KR, Troosters T; PROactive Consortium. Validity of physical activity monitors during daily life in patients with COPD. Eur Respir J. 2013 Nov;42(5):1205-15. doi: 10.1183/09031936.00134312. Epub 2013 Feb 8. PMID 23397303
- [Background] Bosy-Westphal A, Schautz B, Later W, Kehayias JJ, Gallagher D, Muller MJ. What makes a BIA equation unique? Validity of eight-electrode multifrequency BIA to estimate body composition in a healthy adult population. Eur J Clin Nutr. 2013 Jan;67 Suppl 1:S14-21. doi: 10.1038/ejcn.2012.160. PMID 23299866
- [Background] Leelarathna L, Wilmot EG. Flash forward: a review of flash glucose monitoring. Diabet Med. 2018 Apr;35(4):472-482. doi: 10.1111/dme.13584. Epub 2018 Feb 27. PMID 29356072
- [Background] Goodpaster BH, Kelley DE, Thaete FL, He J, Ross R. Skeletal muscle attenuation determined by computed tomography is associated with skeletal muscle lipid content. J Appl Physiol (1985). 2000 Jul;89(1):104-10. doi: 10.1152/jappl.2000.89.1.104. PMID 10904041
- [Background] Martin L, Birdsell L, Macdonald N, Reiman T, Clandinin MT, McCargar LJ, Murphy R, Ghosh S, Sawyer MB, Baracos VE. Cancer cachexia in the age of obesity: skeletal muscle depletion is a powerful prognostic factor, independent of body mass index. J Clin Oncol. 2013 Apr 20;31(12):1539-47. doi: 10.1200/JCO.2012.45.2722. Epub 2013 Mar 25. PMID 23530101
- [Background] Tarnopolsky MA, Pearce E, Smith K, Lach B. Suction-modified Bergstrom muscle biopsy technique: experience with 13,500 procedures. Muscle Nerve. 2011 May;43(5):717-25. doi: 10.1002/mus.21945. Epub 2011 Apr 1. PMID 21462204